CLINICAL TRIAL: NCT03542747
Title: Comparison of the Novel iLTS and Fastrach Intubation Laryngeal Mask for Time to Ventilation in a Simulated Airway.
Brief Title: Comparison of iLTS and LMA Fastrach in a Simulated Airway.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Marc Kriege, MD, MD, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JohannesGUN
Record Dates: First submitted 2018-05-20; First posted 2018-05-31 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Ventilation Therapy; Complications
Keywords: Airway; extraglottic; simulation; laryngeal mask

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time to ventilation with the iLTS (Experimental): Measuring the time to ventilation (ET) based of insert the iLTS until the chest rise of the simulator in seconds
  Interventions: Device: Time to ventilation with the iLTS; Device: Time to ventilation with the Fastrach
- Time to ventilation with the Fastrach (Experimental): Measuring time to ventilation (ET) based of insert the Fastrach until the chest rise of the simulator in seconds
  Interventions: Device: Time to ventilation with the iLTS; Device: Time to ventilation with the Fastrach

INTERVENTIONS:
Device: Time to ventilation with the iLTS — Time to ventilation (ET) based of insert the iLTS until the chest rise of the simulator in seconds
Device: Time to ventilation with the Fastrach — Time to ventilation (ET) based of insert the Fastrach until the chest rise of the simulator in seconds

SUMMARY:
Comparison of time to ventilation based on the chest rising of the Airway Simulator between the iLTS-D and LMA Fastrach

DETAILED DESCRIPTION:
Prior to the study every participant obtained a standardized instruction of each device. In the proposed clinical trial the primary study objective will be to determine whether there is a difference in time to ventilation via endotracheal tube (seconds) for the novel iLTS-D compared to the LMA Fastrach. Time to Ventilation will be defined from when the tip of the extraglottic airway device passed the incisors to the point until confirmation the first chest rise of the high fidelity simulator (Laerdal SimMan). Additionally, two time points before final tracheal placement will evaluated: time to place the EGA and time to ventilate with the EGA after introducing the device into the oral cavity.

ELIGIBILITY:
Inclusion Criteria:

* Medical students
* Present written informed consent of the research participant

Exclusion Criteria:

• inability to consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Time to ventilation via endotracheal tube | 0 to 300 seconds
  time to ventilation will defined from when the Endotracheal tube insert into the extraglottic airway device until the first chest rise

SECONDARY OUTCOMES:
Time to ventilation via extraglottic airway device | 0 to 300 seconds
  time to ventilation will defined from when the device tip passed the incisors to the point until the first chest rise
Intubation attempts | 0 to 300 seconds
  Numbers of successful intubation attempts (1-5 attempts)
Ease of Insertion | 0 to 420 seconds
  Subjective Grading of the insertion process (Lickert Scale from 1 very easy to 5 very difficult)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ott, MD, Study Director — Johannes GU, Mainz
Locations (1):
- Department of Anesthesiology,Prof. C. Werner, Universitätsmedizin of the JG University, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Background] Perkins GD, Olasveengen TM, Maconochie I, Soar J, Wyllie J, Greif R, Lockey A, Semeraro F, Van de Voorde P, Lott C, Monsieurs KG, Nolan JP; European Resuscitation Council. European Resuscitation Council Guidelines for Resuscitation: 2017 update. Resuscitation. 2018 Feb;123:43-50. doi: 10.1016/j.resuscitation.2017.12.007. Epub 2017 Dec 9. No abstract available. PMID 29233740
- [Result] Ott T, Fischer M, Limbach T, Schmidtmann I, Piepho T, Noppens RR. The novel intubating laryngeal tube (iLTS-D) is comparable to the intubating laryngeal mask (Fastrach) - a prospective randomised manikin study. Scand J Trauma Resusc Emerg Med. 2015 Jun 8;23:44. doi: 10.1186/s13049-015-0126-y. PMID 26051498
- [Derived] Ott T, Tschope K, Toenges G, Buggenhagen H, Engelhard K, Kriege M. Does the revised intubating laryngeal tube (ILTS-D2) perform better than the intubating laryngeal mask (Fastrach)? - a randomised simulation research study. BMC Anesthesiol. 2020 May 11;20(1):111. doi: 10.1186/s12871-020-01029-3. PMID 32393169